CLINICAL TRIAL: NCT03617601
Title: Metabolic Equivalent of Task (MET) in the Preoperative Assessment in Aortic Surgery
Status: Completed | Type: Observational
Sponsor: Triemli Hospital (Other)
Responsible Party: Principal Investigator, Alicja Zientara, Resident for cardiac surgery, Triemli Hospital
Other Study IDs: KEK-ZH-Nr: 2017-00801
Record Dates: First submitted 2018-07-06; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Aortic Diseases
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- > 4 MET: Patients with functional capacity over 4 MET
  Interventions: Diagnostic Test: MET
- < 4 MET: Patients with functional capacity under 4 MET
  Interventions: Diagnostic Test: MET

INTERVENTIONS:
Diagnostic Test: MET — Testing of the metabolic equivalent of task before aortic procedure

SUMMARY:
Reliable prediction of the preoperative risk is of crucial importance for patients undergoing vascular operations. The assessment of the metabolic equivalent of task (MET) is an easy clinical evaluation of the functional capacity of an individual. A MET is defined as the resting metabolic rate, that is the amount of the consumed oxygen at rest. According to the MET concept a patient would be considered as "fit for surgery" when the stairs of two flights can be climbed and the housework can be fully managed by oneself.

Hypothesis: Patients with a functional capacity over 4 MET (fit for surgery) have less perioperative complications with the focus on cardiac pathology than patients with less than 4 MET during aortic operations.

Patients and Method: Retrospective analysis of a single center unit of 296 patients undergoing open or endovascular aortic repair.

ELIGIBILITY:
Inclusion Criteria:

* Data of all patients after open and endovascular aortic repair of the descending aorta from May 2009 till March 2016

Exclusion Criteria:

* Data of all patients with isolated operations on the ascending aorta or aortic arch

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 296 patients who received an aortic repair with open or endovascular technique at Triemli Hospital from May 2009 till March 2016
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Survival | up to ten years
  Mean survival during the whole follow up period of both groups, patients with less and more than 4 MET

SECONDARY OUTCOMES:
Perioperative complications | up to 30 days postoperatively
  Complications include perioperative myocardial infarction and stroke, re-operation during first admission (divided in greater and smaller re-operations)
Coronary artery bypass grafting, percutaneous coronary intervention/Stenting | up to ten years
  Interventions including revascularisation or other kind of heart surgery or treatment because of cardiac pathology

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Attigah, MD, Study Chair — Triemli Hospital Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zientara A, Schwegler I, Dzemali O, Bruijnen H, Bernheim A, Dick F, Attigah N. Evaluation of metabolic equivalents of task (METs) in the preoperative assessment in aortic repair. BMC Surg. 2021 Mar 13;21(1):130. doi: 10.1186/s12893-021-01143-0. PMID 33714271